CLINICAL TRIAL: NCT04008342
Title: Effectiveness of a Multisensory Stimulation Intervention on Neuropsychiatric Symptoms in Moderate to Advanced Dementia: a Randomized Controlled Clinical Trial
Brief Title: Multisensory Stimulation in Dementia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Paulo Caramelli, Professor of Neurology, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Paulo Caramelli
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Dementia
Keywords: aged; nonpharmacological intervention; multisensory stimulation; neuropsychiatric symptoms; long-term care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: An experimental pre- and postintervention design was used. The participants were recruited from philanthropic LTC institutions for aged people and allocated in experimental group and control group.
Who Masked: Outcomes Assessor
Masking Description: The evaluations were performed by a blind investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group (IG) was submitted to 16 multisensory sessions that followed the protocol.
  Interventions: Other: Multisensory intervention
- Control group (No Intervention): The control group (CG) received usual care with routine interventions and services in the LTC, such as bath, hygiene care, watching TV and so on.

INTERVENTIONS:
Other: Multisensory intervention — The intervention group (IG) was submitted to 16 individual multisensory stimulation sessions that followed the protocol. In each session, at least two senses are stimulated in a safe, quiet and confidential environment. The sessions lasted 30 minutes and were conducted twice a week, on the same day and time whenever possible. Nonetheless, the session could be interrupted when the participant wished or if the therapist observed that the patient was uncomfortable. A nondirective approach and one-to-one intervention were adopted.
  Arms: Intervention group

SUMMARY:
Dementia is one of the main causes of disability in the elderly. It is characterized by cognitive, functional and social impairment, as well as behavioral changes. Neuropsychiatric symptoms (NPS) are experienced by patients and observed by caregivers during the natural course of dementia. These symptoms, such as apathy, depression and agitation, are a heterogeneous group of noncognitive symptoms and behaviors. When these symptoms are present, it is more likely that the elderly will be institutionalized as the caregivers will be overloaded with demands. Pharmacological treatment presents little efficacy for the adequate control of these symptoms, and nonpharmacological interventions have been recommended as the first line of treatment. Multisensory stimulation (MSS), a nonpharmacological intervention, is one of the possibilities for intervention in people with dementia and NPS. MSS aims to stimulate the five primary senses, namely, hearing, sight, taste, smell and touch, through pleasurable sensory experiences, in a safe and relaxed environment. This work aims to investigate the effects of an MSS protocol in aged people with dementia living in long-term care institutions in Brazil.

DETAILED DESCRIPTION:
Background: Neuropsychiatric symptoms (NPS) in people with dementia frequently evolve with progression of the disorder. Nonpharmacological interventions are the first-line treatment to control NPS in dementia. Multisensory stimulation (MSS) is a nonpharmacological intervention that is conducted by stimulating one or more of the five senses of the body with pleasant sensory experiences. This work aims to investigate the effects of a MSS protocol in elderly people with moderate to advanced dementia living in long-term care institutions in Brazil.

Methods: A specific MSS protocol was developed by the researchers for the study. Sixty elderly people with moderate to advanced dementia (Clinical Dementia Rating of 2 or 3 and a Mini-Mental State Examination score ≤17) were randomly allocated to intervention (n=30) and control (n=30) groups. The sample size estimation was established with a paired bilateral t-test with a 0.05 significance level. This sample size would have 80% power to detect a mean difference of 9.50 in the NPI scores from pre- to post-intervention and a standard deviation of 17.28, as proposed by Fu et al. (2013). The intervention group participated in 16 individual 30-minute sessions over eight weeks in a quiet room, and the control group received usual care.

The MSS program includes eight sessions. During these sessions, the five body senses (sight, taste, hearing, smell, and feeling) are stimulated using songs, fruits, fiber optic lamps, natural scents, among other stimuli, to promote interactions between the participants and the therapist, as well as the objects. In each session, at least two senses are stimulated in a safe, quiet and confidential environment. The sessions last 30 minutes and are conducted twice a week, on the same day and time whenever possible. Nonetheless, the session can be interrupted when the participant wishes or if the therapist observes that the patient is uncomfortable. A nondirective approach and one-to-one intervention were adopted.The MSS protocol was conducted by an occupational therapist. In this study, the eight-session protocol was used twice, that is, the protocol was repeated from the ninth session forward, but the protocol was customized for each participant by consideration of the participants' interests in previous sessions and the protocol rules.

ELIGIBILITY:
Inclusion Criteria residents:

* elderly person;
* moderate or advanced dementia diagnosis (Clinical Dementia Rating (CDR) of 2 or 3);
* score equal to or less than 17 on the Mini-Mental State Examination;

Inclusion Criteria caregivers:

* Formal caregivers involved in the direct care of these elderly patients;
* Formal caregivers did not have holidays during the intervention period.

Exclusion Criteria:

* profound vision and hearing loss;
* presence of any additional psychiatric or neurological diagnosis (e.g., schizophrenia or intellectual disability);
* plan to relocate to another residence in less than three months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Effects on agitation | 10-20 minutes
  To measure agitation, the Cohen-Mansfield Agitation Inventory (CMAI) was used. The maximum score was 144 points and a higher score indicated more frequent symptoms
Effects on neuropsychiatric symptoms | 10-20 minutes
  The frequency and intensity of neuropsychiatric symptoms (NPS) were assessed by the Neuropsychiatric Inventory (NPI). The scale considered 12 domains and the total score (0-144) was calculated by multiplying the frequency (1-4) and the severiity (1-3) of the symptoms. A higher score indicated more severe NPS. Assessment results are presented for the total score and the four neuropsychiatric subsyndromes of the NPI: hyperactivity, psychosis, affective symptoms and apathy.
Effects on depression | 10-20 minutes
  The Cornell Scale for Depression in Dementia (CSDD) was employed to evaluate depressive symptoms. Each item was scored as zero (absent), one (mild), two (severe), or unable to evaluate, and the total score (0-38) was calculated by adding the item scores. The scale is divided into five subscales: mood-related signs, behavioral disturbance, physical signs, cyclic functions and ideational disturbance. The total score ranged from 0 to 38; a higher score indicated greater levels of depression.
Effects on apathy | 5-10 minutes
  The Apathy Scale (AS) was used as a measure of apathy symptoms. The maximum score was 42 points, and higher scores indicated greater intensity of these symptoms

SECONDARY OUTCOMES:
Effect on functional status | 10-20 minutes
  The Barthel Index was used to assess functional independence and mobility in daily life activities. The total score ranged from 0-100 points, and higher scores indicated more independence.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa S Serelli, PhD, Principal Investigator — Federal University of Minas Gerais; Marcella G Assis, PhD, Principal Investigator — Federal University of Minas Gerais; Paulo Caramelli, MD, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- School of Medicine, Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No